CLINICAL TRIAL: NCT04445350
Title: Motor Learning in Knee Osteoarthritis Therapy - A New Rehabilitation Approach
Brief Title: Motor Learning in Knee Osteoarthritis
Acronym: MLKOA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Pölten University of Applied Sciences (Other)
Collaborators: Danube University Krems (Other); Karl Landsteiner University of Health Sciences (Other); Orthopedic Hospital Speising (Unknown)
Responsible Party: Principal Investigator, Wondrasch, FH-Professor Barbara Wondrasch, PhD, St. Pölten University of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: StPoltenUAS
Record Dates: First submitted 2020-06-09; First posted 2020-06-24 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Knee Osteoarthritis; Lower Extremity Biomechanics; Physiotherapy
Keywords: Physiotherapy; External Focus Of Attention; Knee Adduction Moment; Gait Analysis; Osteoarthritis; Motor Learning
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External focus of attention training program (Experimental): The intervention group receives a strength and neuromuscular training program. The training instructions have an external focus of attention.
  Interventions: Other: External Focus Of Attention
- Internal focus of attention training program (Active Comparator): The control group receives a strength and neuromuscular training program. The training instructions have an internal focus of attention.
  Interventions: Other: Internal Focus Of Attention

INTERVENTIONS:
Other: External Focus Of Attention — Instructions and feedback are used to direct the learner's focus to an external source (e.g. the effect the intended movement has) promoting long-term learning by stimulating automatic cognitive control processes.
  Arms: External focus of attention training program
Other: Internal Focus Of Attention — In contrast, adopting an internal focus of attention (e.g. focus on specific body areal) can disrupt automatic control processes and interfere automatic movement.
  Arms: Internal focus of attention training program

SUMMARY:
Non-surgical treatment options, like exercise therapy, show excellent short-term effects regarding pain reduction and improvement of knee function. However, mid- and long-term effects are missing so far. This might indicate that long-lasting changes in motor-skill performance (Motor Learning) have not occurred. Motor learning is associated with permanent changes in the capability for skilled movement behavior avoiding unfavorable joint loads and inappropriate muscle activation patterns, leading to compensatory movement strategies. One-sided and high repetitive loads in the knee joint could be one reason for the progression of knee osteoarthritis. Physiotherapeutic strategies should therefore be able to stimulate motor learning processes. In physiotherapy, motor learning can be optimized by using instructions and feedback, targeting an external focus of attention, when learning specific movement patterns. This study investigates the effects of a 12 week exercise therapy program, using an external focus of attention, on functional and biomechanical parameters in patients with knee osteoarthritis. To measure possible changes, functional measurements are taking place at baseline, after 6, 12 and 24 weeks. The biomechanical measurements (3D gait analysis) are taking place at baseline, after 12 and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Kellgren-Lawrence-Score 1-3
* BMI < 33
* Free range of motion in the knee joint

Exclusion Criteria:

* Activated knee osteoarthritis
* Lower extremity surgery in the past 6 weeks
* Intake or injection of corticosteroids in the past 3 month
* Long-term medication non-steroidal anti-inflammatory drugs
* Neurological diseases
* Drug or alcohol abuse

Ages: 45 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-04-30 (Estimated)

PRIMARY OUTCOMES:
Knee Adduction Moment (change over a period of 6 month with 3 measurement dates) | Baseline, 12 weeks, 24 weeks
  3D gait analysis during walking
Knee Osteoarthritis Outcome Score (change over a period of 6 month with 4 measurement dates) | Baseline, 6 weeks, 12 weeks, 24 weeks
  Questionnaire; Minimum value: 0 (highest limitation), Maximum: 100 (no limitation)
Star Excursion Balance Test (change over a period of 6 month with 4 measurement dates) | Baseline, 6 weeks, 12 weeks, 24 weeks
  An established test to determine movement control and balance ability. The test person stands on one leg and will is asked to stretch the non supporting leg as far as possible in the directions presented.
Isometric strength tests (change over a period of 6 month with 4 measurement dates) | Baseline, 6 weeks, 12 weeks, 24 weeks
  Measures the isometric force of the knee extensors, knee flexors, hip abductors, hip extensors and hip external rotators with a portable dynamometer
Six minute walking test (change over a period of 6 month with 4 measurement dates) | Baseline, 6 weeks, 12 weeks, 24 weeks
  The six minute walking test is a reliable measuring tool to examine the distance a person can walk in a given time period.

CONTACTS AND LOCATIONS:
Locations (1):
- Sankt Pölten University of Applied Sciences, Sankt Pölten, Lower Austria, Austria